CLINICAL TRIAL: NCT01959061
Title: Raltitrexed and Oxaliplatin and Lipiodol Transcatheter Arterial Chemoembolization for Advanced Colorectal Cancer
Brief Title: Efficacy and Safety of Raltitrexed-based Transarterial Chemoembolisation(TACE)for Colorectal Cancer Liver Metastases
Acronym: TACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCTTQ-01
Record Dates: First submitted 2013-09-18; First posted 2013-10-09 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Advanced colorectal cancer of liver metastatic
MeSH Terms: interventions — raltitrexed; Oxaliplatin; Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltitrexed and Oxaliplatin (Experimental): Raltitrexed and Oxaliplatin were mixed with 10-15 ml lipiodol by arterial chemoembolization on day 1 and during each 28-day cycle.
  Interventions: Drug: Raltitrexed; Drug: Oxaliplatin; Drug: lipiodol

INTERVENTIONS:
Drug: Raltitrexed — 4mg, every 4 weeks,transhepatic arterial infusion
Drug: Oxaliplatin — 100~150mg, every 4 weeks, transhepatic arterial infusion
Drug: lipiodol — 5-20ml, every 4 weeks, hepatic artery embolization

SUMMARY:
To evaluate the efficacy and safety of Raltitrexed for advanced colorectal cancer

DETAILED DESCRIPTION:
evaluate the efficacy and safety of Raltitrexed and oxaliplatin and lipiodol transcatheter arthrial chemoembolization for in refractory colorectal carcinoma with liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal adenocarcinoma
2. Disease limited to the liver Unresectable disease by surgery or other local therapies
3. Age >18 years
4. ECOG performance status 0-2,Child pugh A or B
5. Expected survival ≥ 3 months
6. Adequate hematological, hepatic, and renal function

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with severe organ dysfunction or failure
3. With severe cardiovascular disease, or mental
4. Extraliver metastases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survivial | 8 months after last patient randomized
  From date of randomization until date of first documented PD, date of death

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Wang, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided